CLINICAL TRIAL: NCT06334302
Title: The Effect of Omega Galil Hazelnut Chocolate Spread "O'Sweet Spread" With 80% Reduced Sucrose on Glucose Response of People With TID - a Randomized, Double-blind, Active Control Trial
Brief Title: The Effect of Omega Galil Hazelnut Chocolate Spread "O'Sweet Spread" With 80% Reduced Sucrose on Glucose Response of People With TID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Omega 3 Galilee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: RMC0362-23ctil
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Type1diabetes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega Galil O'Sweet hazelnut cocoa spread (Experimental): Omega Galil O'Sweet hazelnut cocoa spread is composed of 8% sucrose, 26% MCT oil, 6% cocoa butter, 6% cocoa powder, 10% Hazelnut paste, 24% fibers, 13% rice flour. It contains a total of 27.3 gram carbohydrates/ 100gram, 520 kcals/100 grams, and very low estimated GL according to healthy adults
  Interventions: Other: Omega Galil Hazelnut Chocolate Spread "O'Sweet Spread"
- Nutella hazelnut cocoa spread (Active Comparator): Nutella hazelnut cocoa spread is composed of 56% sugar, 30% vegetable fat, 13% Hazelnut paste, milk powder (8.7%), and cocoa powder (7.4%), containing a total of 57.5 grams carbohydrates /100grams, 532 kcals/100 grams, and an estimated GL of 4
  Interventions: Other: Active Control-Nutella hazelnut cocoa spread

INTERVENTIONS:
Other: Omega Galil Hazelnut Chocolate Spread "O'Sweet Spread" — Omega Galil O'Sweet hazelnut cocoa spread is composed of 8% sucrose, 26% MCT oil, 6% cocoa butter, 6% cocoa powder, 10% Hazelnut paste, 24% fibers, 13% rice flour. It contains a total of 27.3 gram carbohydrates/ 100gram, 520 kcals/100 grams, and very low estimated GL according to healthy adults
  Other Names: "O'Sweet Spread"
  Arms: Omega Galil O'Sweet hazelnut cocoa spread
Other: Active Control-Nutella hazelnut cocoa spread — Nutella hazelnut cocoa spread is composed of 56% sugar, 30% vegetable fat, 13% Hazelnut paste, milk powder (8.7%), and cocoa powder (7.4%), containing a total of 57.5 grams carbohydrates /100grams, 532 kcals/100 grams, and an estimated GL of 4
  Other Names: Nutella hazelnut cocoa spread
  Arms: Nutella hazelnut cocoa spread

SUMMARY:
Omega Galil has developed a novel fatty sweetener that allows the use of up to 80% less sugar (particularly sucrose) and yet achieves a natural sweet flavor, using a novel technology of milling the natural sucrose crystals together with oil and thus creating a micro-suspension of sugar in oil or fat. The suspension increases the surface area of the sugar particles and thus a lower quantity of sugar is required in order to reach an enhanced perception of sweetness at the sweet taste receptors in the mouth. Omega Galil provides fatty food products that use up to 80% less sucrose, while tasting as sweet as regular sugar sweetened foods, with no aftertastes of sugar substitutes, and no chemical modifications or additives.

Postprandial glucose (PPG) excursions in Type 1 Diabetes happen mainly due to a delay in subcutaneous insulin absorption and action, but also among other factors, depend on the meal composition. The glycemic index (GI) ranks foods based on acute glycemic response over a 2-h period of 50 g of available carbohydrates (CHO) of a test food compared with the reference standard glucose. Glycemic Load (GL) is a GI-weighted measure of carbohydrate content, which estimates the impact of carbohydrate intake using the GI while taking into account the amount of carbohydrates that are eaten in a serving. Several studies have demonstrated differences in PPG after consumption of low versus high GI meals, with rapid glucose spikes following high GI meals . Helping people with T1D achieve a diet with a lower glycemic load can improve both their quality of life and their diabetes-associated complications.

The proposed randomized, double blind, cross-over, active control, clinical trial aims to:

1. compare the glycemic response of T1D subjects to 20 grams of the O'Sweet sugar-reduced spread containing 8% sugar and a total of 1.6 grams of sucrose per meal, with their glycemic response to 20 grams of control Nutella spread, containing 56% sugar and a total of 11 grams sucrose per meal.
2. compare the acceptance ("Not sweet enough, just right or too sweet") Labeled Magnitude score of O'Sweet compared to the control spread (Nutella).

ELIGIBILITY:
Inclusion Criteria:

* T1D patients with diabetes duration >1 year
* 18-35 years of age
* Normal weight (BMI 20- 30 kg/m2)
* Non-smoker
* Hemoglobin A1C <9%
* Patient treated with Continuous Glucose Monitoring system (CGM's)

Exclusion Criteria:

* Acute Upper Respiratory Tract Infection (URTI) within 2 weeks of enrollment
* A gastro-intestinal condition that could disrupt intestinal absorption or motility, and thereby impair postprandial glucose absorption (e.g. diabetic gastroparesis, celiac disease, or malabsorption).
* A chronic illness in the past 5 years, including among others inflammatory, metabolic, neoplastic, and congenital disease.
* Use of medications other than insulin (e.g. Antibiotics/antifungal, analgesics) during the study and 2 weeks before enrollment;
* Neuro-psychiatric disorders
* Known food allergies or intolerances
* Self-reported sinus, taste or smell dysfunction
* Pregnant or lactating women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-04-25 (Estimated)

PRIMARY OUTCOMES:
Delta postprandial glucose level | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  The difference between pre-meal and peak postprandial glucose level in each of the two 2 hours' meal tests.

SECONDARY OUTCOMES:
Incremental area under the curve (iAUC) | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  Incremental area under the curve (iAUC) using continuous glucose sensor data > 180 mg/dl between the beginning of the meal and 2 hours postprandial (defined as the postprandial period).
Peak postprandial glucose level | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  The peak postprandial glucose level during the 2-hour postprandial period
Time in range (TIR) of 70-180 mg/dl | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  Time in range (TIR) of 70-180 mg/dl during the postprandial period
Percentage of subjects who reached the desired glucose target | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  The percentage of subjects who reached the desired glucose target (70-180 mg/dl) during the postprandial period (70% of the time)
The percentage of time spent above 180 mg/dl | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  The percentage of time spent above 180 mg/dl
The percentage of time spent above 250 mg/dl | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  The percentage of time spent above 250 mg/dl
The percentage of time spent above 350 md/dl | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  The percentage of time spent above 350 md/dl
Labeled Magnitude Scale (gLMS) | first meal teat visit 1 (day 1) and second meal test visit 2 (2 weeks)
  Acceptance of the sweetness level Labeled Magnitude Scale (gLMS)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Gavan, PHd, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No